CLINICAL TRIAL: NCT05527366
Title: The Effect of Auricular Vagus Stimulating on Pain, Disability and Sleep in Non Specific Chronic Neck Pain
Brief Title: Effect of Auricular Vagus Stimulating in Non Specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Vagus; Autonomic Nervous System
MeSH Terms: conditions — Neck Pain | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Conservative treatment
  Interventions: Other: Vagus stimulation
- Vagus Stimulation Group (Experimental): Vagus Stimulation Group
  Interventions: Other: Consevative treatment

INTERVENTIONS:
Other: Vagus stimulation — The Vagus Stimulation Group received auricular vagus stimulation for a total of 15 sessions of 25 minutes 5 days a week. The patients were applied with vagustim device consisting of TENS device with electrodes placed bilaterally in the outer ear with headphones that can be selected according to ear size. During the application, the gel was used to avoid causing any damage and to ensure conductivity. It is placed so that tragus and konkaya are facing. The pulse duration of the TENS device is less than 500 microseconds, the frequency is 10 Herzt, the module was applied in TENS mode and in the form of a biphasic asymmetric wave.
  Arms: Control Group
Other: Consevative treatment — A total of 15 sessions 5 days a week, 20 minutes of hotpack, 20 minutes of TENS, 5 minutes of 1,3 watt/cm2 ultrasound consisting of a total of 25 minutes of treatment was applied to the neck area.
  Arms: Vagus Stimulation Group

SUMMARY:
The aim of our study is to compare the efects of conventional treatment and vagus nerve stimulation on pain, normal joint movement, disability and sleep in non-specific chronic neck pain.

36 patients aged between 18 and 65 years with non-specific neck pain participated in our randomly planned study. All these patients were divided into 2 groups. Demographic and physical characteristics of the patients were recorded. The first group was treated with auricular vagus nerve stimulation. Conservatire treatment that consists of hotpack, transcutaneous electrical nerve stimulation (TENS) and therapeutic ultrasound was applied to the second group. In addition to their treatment, some home exercises were given and tought. Pain was assessed with a visual analog scale (VAS). Muscle strength was evalvated with a digital hand dynamometer. Neck normal joınt motion was evaluated with goniometer clinometer which is a mobile phone application. While disability was mensured with the neck disability index, sleep quality was evalvated with the Pittsburg sleep questionnaire. All the measurements were recorded before the trearment and after the 15 session treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* people with non-specific neck pain

Exclusion Criteria:

* Who has neurological problems,
* who has vision and hearing loss,
* who has a tumor and infection in the cervical region,
* who has undergone surgery related to the cervical region,
* who has had a cervical streroid injection in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 3-week change in pain intensity
  Pain severity Within the scope of this study, a Visual Analog Scale was applied, with both ends marked between 0 and 10, 100 mm long and marked every 10 mm; the patient was marked according to his own pain level, scored between 0-10. Deciphered. Deciphered. The Visual Analogue Scale was applied. 0 was rated as "no pain" and 10 as "unbearable level of pain"
Muscle strength Measurement | 3-week change in muscle strength
  Muscle strength was measured with La Fayette brand digital hand dynamometer. Flexion, extension, right and left lateral flexion of the neck were measured with the device. The patients were fixed to the stretcher with T3 and spina iliac superior ventro tapes. Each movement measurement was repeated 3 times at December intervals of 15 seconds
Joint Range of Motion Measurement | 3-week change in Range of motion
  Neck region flexion, extension, right and left lateral flexion joint range of motion was evaluated by climatometer. The tests were performed in a back-supported chair. While the phone application called Goniometer was open, the evaluation was performed by placing it in a vertical position in front of the ear for flexion and extension measurements, and by placing the measurement line on the side that was not measured so as not to prevent movement in lateral flexion measurements, so that the measurement line was flush with the eyes. Rotation movements were measured by placing the phone on the person's head to follow the nose alignment. The ROM value was taken as the average of the 3 active movement spans made by the individuals after the movement made passively once by the physiotherapist.
Assessment of dysability | 3-week change in dysability
  The level of chronic neck pain affecting daily life activities was assessed by the Neck Disability Index (NDI). The validity of this index in Turkish was made by Telci et al. Neck Disability Index consists of 10 items and Article 4 of subjective symptoms (pain intensity, headache, concentration, sleep) substance other 6 activities of daily living (personal care, lifting, reading, business, car handling and leisure pursuits) is related to.The classification of disability according to neck disability index score is as follows; 0-4: no disability, 5-14: mild disability, 15-24: moderate disability, 25-34: severe disability, >34: full disability.
Evaluation of sleep quality | 3-week change in sleep quality
  Pittsburgh sleep quality index, Agargün et al. it is turkified by. The index is a 19-item self-report that evaluates sleep disturbance and quality in the last one-month period. it consists of 24 questions, 19 questions are self-report questions, 5 questions are answered by a spouse or roommate. The 18 scored questions of the scale consist of 7 components. These are subjective sleep quality, sleep duration, sleep latency, sleep disturbance, habitual sleep activity, use of sleeping pills, and daytime dysfunction.The global score obtained ranges from 0-21, and high values indicate that the quality of sleep is poor Decently, the level of sleep disturbance is high. A global score of 5 or above indicates that the quality of sleep is clinically significantly poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No